CLINICAL TRIAL: NCT01384396
Title: A Clinical Study of KW-3357 in Patients Diagnosed as Disseminated Intravascular Coagulation (DIC) by the Diagnostic Criteria for DIC Established by the Japanese Ministry of Health and Welfare
Brief Title: A Clinical Study of KW-3357 in Patients With DIC
Acronym: 3357-005
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kyowa Kirin Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3357-005
Record Dates: First submitted 2011-06-27; First posted 2011-06-29 (Estimated); Last update posted 2017-03-24 (Actual); Status verified 2017-03

CONDITIONS: Disseminated Intravascular Coagulation (DIC)
MeSH Terms: conditions — Disseminated Intravascular Coagulation

ARMS (1):
- KW-3357 (Experimental)
  Interventions: Drug: KW-3357

INTERVENTIONS:
Drug: KW-3357 — Intravenous infusion once a day

SUMMARY:
To evaluate the efficacy and safety of KW-3357 with concomitant use of heparin using multi-center, non-comparative, open-label method in patients diagnosed as disseminated intravascular coagulation (DIC) by the diagnostic criteria for DIC established by the Japanese Ministry of Health and Welfare.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed or suspected as DIC by the diagnostic criteria for DIC established by the Japanese Ministry of Health and Welfare
* Antithrombin activity <= 70%
* Written informed consent from patient or guardian

Exclusion Criteria:

* Anamnesis or complication of serious drug allergy
* Serious liver disorder, such as fulminant hepatitis and decompensated cirrhosis
* Pregnant, nursing, or possibly pregnant woman
* Possibility for the promotion of bleeding by concomitant use of heparin

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2011-12; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Safety | up to 6 days (or discontinuation)
  Number of patients with adverse events
DIC resolution | 6 days (or discontinuation)
  Resolution from DIC by the diagnostic criteria for DIC established by the Japanese Ministry of Health and Welfare

SECONDARY OUTCOMES:
DIC score | Screening, 2, 3, 4, 5, 6 days (or discontinuation)
  Based on the diagnostic criteria for DIC established by the Japanese Ministry of Health and Welfare
Mortality | 28 days
Plasma antithrombin activity | Screening, 2, 3, 4, 5, 6 days (or discontinuation)

CONTACTS AND LOCATIONS:
Locations (1):
- Kanazawa, Japan